CLINICAL TRIAL: NCT07244640
Title: Clinical Study on Non-Invasive Fundus Retinal Detection Technology for Early Diagnosis of Parkinson's Disease
Brief Title: Non-Invasive Fundus Retinal Detection Technology for Early Diagnosis of Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: College of Optical Science and Engineering, Zhejiang University (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20251675
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Parkinson's Disease: Patients who meet the 2015 International Movement Disorder Society clinical diagnostic criteria for Parkinson's disease, with a Hoehn and Yahr stage of 1 to 2.5 and a disease duration of ≤5 years.
  Interventions: Diagnostic Test: non-invasive fundus retinal detection
- Parkinson's Syndromes: Patients who meet the International Movement Disorder Society diagnostic criteria for atypical parkinson's syndromes (including progressive supranuclear palsy, dementia with Lewy bodies, and corticobasal degeneration), multiple system atrophy (P subtype), or secondary parkinson's syndrome (drug-induced: having taken antipsychotic medications for ≥3 months; vascular: confirmed by brain MRI showing leukoaraiosis/lacunar infarction), with a disease duration of ≤5 years.
  Interventions: Diagnostic Test: non-invasive fundus retinal detection
- Essential Tremor: Patients who meet the 2018 International Movement Disorder Society clinical diagnostic criteria for essential tremor, with no parkinsonian symptoms, and a disease duration of ≥1 year.
  Interventions: Diagnostic Test: non-invasive fundus retinal detection
- Healthy Control: Individuals with no parkinsonian symptoms (confirmed by neurological examination) and no use of antipsychotic/dopaminergic medications in the past 3 months.
  Interventions: Diagnostic Test: non-invasive fundus retinal detection

INTERVENTIONS:
Diagnostic Test: non-invasive fundus retinal detection — functional optical coherence tomography angiography-retinal neurovascular coupling (fOCTA-rNVC) detection technology

SUMMARY:
The objective of this observational study is to investigate whether non-invasive fundus retinal detection technology can be used for the early diagnosis of parkinson's disease (PD). It aims to answer the following primary questions: the sensitivity and specificity of non-invasive fundus retinal detection technology in the early diagnosis of PD; and whether this technology offers advantages over dopamine transporter positron emission tomography (DAT-PET), a conventional screening method for PD. The researchers will analyze the diagnostic performance of this technology for early-stage PD patients among cohorts including early parkinson's disease, parkinson's syndromes, essential tremor patients, and healthy individuals. Furthermore, in PD patients who concurrently undergo DAT-PET imaging, the study will compare the diagnostic value of non-invasive retinal imaging against that of DAT-PET.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 40-80 years; 2. Parkinson's Disease Group: Patients who meet the 2015 International Movement Disorder Society clinical diagnostic criteria for Parkinson's disease, with a Hoehn and Yahr stage of 1 to 2.5 and a disease duration of ≤5 years; 3. Parkinson's Syndromes Group: Patients who meet the International Movement Disorder Society diagnostic criteria for atypical parkinson's syndromes (including progressive supranuclear palsy, dementia with Lewy bodies, and corticobasal degeneration), multiple system atrophy (P subtype), or secondary parkinson's syndrome (drug-induced: having taken antipsychotic medications for ≥3 months; vascular: confirmed by brain MRI showing leukoaraiosis/lacunar infarction), with a disease duration of ≤5 years; 4. Essential Tremor Group: Patients who meet the 2018 International Movement Disorder Society clinical diagnostic criteria for essential tremor, with no parkinsonian symptoms, and a disease duration of ≥1 year; 5. Healthy Control Group: Individuals with no parkinsonian symptoms (confirmed by neurological examination) and no use of antipsychotic/dopaminergic medications in the past 3 months; 6. All subjects have provided written informed consent and are willing to comply with the study procedures.

Exclusion Criteria:

* 1. Presence of severe ocular fundus diseases, such as glaucoma, cataract, retinal detachment, macular degeneration, etc; 2. Inability to tolerate the non-invasive fundus retinal detection; 3. Known allergy or investigator-suspected high risk of allergy to anti-PD drugs; 4. Presence of severe cardiovascular or cerebrovascular diseases (e.g., coronary heart disease, myocardial infarction, stroke, etc.), hepatic or renal dysfunction, cancer, or other conditions that may affect the prognosis; 5. Pregnancy or lactation; 6. Presence of active infectious diseases (e.g., tuberculosis, AIDS) or systemic inflammatory diseases (e.g., rheumatoid arthritis); 7. Presence of psychiatric disorders.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll four distinct groups: (1)patients who meet the 2015 International Movement Disorder Society clinical diagnostic criteria for Parkinson's disease, with a Hoehn and Yahr stage of 1 to 2.5 and a disease duration of ≤5 years; (2)patients with Parkinson's syndromes meeting respective MDS criteria; (3) patients with essential tremor meeting the 2018 MDS clinical diagnostic criteria; and (4) healthy controls. Detailed inclusion and exclusion criteria are listed in Eligibility Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of non-invasive fundus retinal detection technology for early parkinson's disease diagnosis | At enrollment
  Sensitivity and specificity will be calculated by comparing the results of non-invasive fundus retinal detection against the clinical diagnostic criteria. Values with 95% confidence intervals will be reported.
Area under the ROC curve (AUC) of retinal parameters for discriminating early parkinson's disease | At enrollment
  The AUC will be computed to evaluate the overall discriminatory power of continuous retinal parameters.

SECONDARY OUTCOMES:
Differential diagnostic accuracy of non-invasive fundus retinal detection technology | At enrollment
  To evaluate the ability of non-invasive fundus retinal detection technology in differentiating among patients with early parkinson's disease, parkinson's syndromes, and essential tremor. Accuracy will be calculated based on the proportion of patients correctly classified into their clinical diagnostic groups (as defined by the international MDS criteria) using retinal parameters.
Comparison of diagnostic accuracy between non-invasive fundus retinal detection technology and DAT-PET in early parkinson's disease | At enrollment
  To evaluate and compare the capability of non-invasive fundus retinal detection technology and dopamine transporter positron emission tomography (DAT-PET) in diagnosing early parkinson's disease, against the clinical diagnostic criteria. Metrics including sensitivity, specificity, AUC, and agreement (e.g., Kappa) will be assessed and compared between the two methods.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China